CLINICAL TRIAL: NCT04230603
Title: Tissue Characterisation With Hyperspectral Imaging Methods
Brief Title: Tissue Characterization With Hyperspectral Imaging (HSI)
Acronym: HSIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Dr. Boris Jansen-Winkeln, Boris Jansen-Winkeln, University of Leipzig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201905
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Tissue Perfusion; Tumor; Inflammation; Inflammatory Bowel Diseases
Keywords: hyperspectral imaging; tissue detection; tumor detection; infammatory bowel disease; colorectal cancer
MeSH Terms: conditions — Neoplasms; Inflammation; Inflammatory Bowel Diseases; Colorectal Neoplasms | interventions — Hyperspectral Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyperspectral imaging (Experimental): diagnostic hyperspectral imaging of the human tissue an correlation with local blood parameters and local pathological examination
  Interventions: Procedure: Hyperspectral imaging; Diagnostic Test: Lactate acid measurement; Diagnostic Test: pathological examination

INTERVENTIONS:
Procedure: Hyperspectral imaging — Photos were taken with the hyperspectral camera of the human tissue
  Other Names: Marking of the target region (Suture/Clip/ink)
Diagnostic Test: Lactate acid measurement — At the marked regions of the specimen, a lactate acid measurement was performed.
Diagnostic Test: pathological examination — At the marked regions of the specimen, the pathological examination was performed.

SUMMARY:
Hyperspectral Imaging (HSI) is a contact free method to analyse the from the tissue reflected light in the range of 500-1000nm. Aim of the study is to identify special reflex patterns to identify special tissue

DETAILED DESCRIPTION:
This HSI-camera provides hyperspectral images with a high spectral resolution (5 nm) in the visible and near infrared range (500-1000 nm). A RGB image and 4 false color images that represent physiologic parameters are intraoperatively provided by an analysis software. But after the procedure all spectral datasets could be investigated. To analyse and differentiate the different tissues, a catalog database is needed of all tissues including Tumors.

ELIGIBILITY:
Inclusion Criteria:

* All patients with surgical procedure

Exclusion Criteria:

* inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-01-02 (Estimated); Study Completion 2022-06-02 (Estimated)

PRIMARY OUTCOMES:
Tumor detection with HSI | direct during the Operation (ca. 15-20 Minutes)
  Due to the non-invasive diagnostics with the HSI camera, tumor tissue can be distinguished from healthy tissue.
Tissue recognition with HSI | after the operation within 24 hours
  different tissues can be differentiated from each other with HSI
Inflammatory classification with HSI | after the operation within 24 hours
  Classification of the grade of the inflammation e.g. in IBD

SECONDARY OUTCOMES:
Tissue perfusion | direct during the Operation (ca. 10-15 Minutes)
  Tissue perfusion in the upper and lower tissue layers measured with the HSI Camera

CONTACTS AND LOCATIONS:
Overall Officials: Ines Gockel, MD, Prof., Study Director — University of Leipzig
Locations (1):
- Universitätsklinikum Leipzig - AöR, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
no sharing